CLINICAL TRIAL: NCT05085847
Title: Molecular and Epigenetic Mechanisms Underlying Cognition Functions and Stress Response: Mindfulness-based Intervention
Brief Title: Effects of Mindfulness-based Intervention on Epigenetic Mechanisms, Cognition Function, Stress Response, and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Flávia Marçal Pessoa, Co-investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3.159.669
Record Dates: First submitted 2021-06-17; First posted 2021-10-20 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Mindfulness; DNA Methylation; Learning and Memory; Stress; Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention (MBI) (Experimental): Participants received mindfulness training for 8 weeks (two-hour meetings; 16 hours total)
  Interventions: Other: Mindfulness meditation training
- Active control group (Active Comparator): Participants received lectures for 8 weeks (two-hour meetings; 16 hours total)
  Interventions: Other: Active control

INTERVENTIONS:
Other: Mindfulness meditation training — Mindfulness-based intervention encompasses different practices which intend to exercise awareness by using mindfulness meditation training moment by moment. Thus, practices such as mindful breathing, compassionate communication, loving-kindness, self-compassion, mindful listening, dealing with difficulties, the 3 step meditation, walking meditation, body scan with progressive relaxation, thoughts, emotions, gratitude, and sounds and breathing will be teaching to participants. Mindfulness training will be conduct by two instructors with more than 30 years' experience in meditation practices (Zen and Tibetan Buddhist approach to mind-training) and extensive mindfulness teaching and practices (> 5 years each) experiences.
  Arms: Mindfulness-based intervention (MBI)
Other: Active control — Participants will receive lectures that provide cognitive and sensorial stimulus which does not specifically involve awareness training (meditation). Lesson topics include science.
  Arms: Active control group

SUMMARY:
The purpose of this study is to assess the effect of a mindfulness-based intervention on DNAmethylation, cognitive functions, stress response, and well-being in healthy female adults.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all volunteers giving written informed consent will undergo a 1-3 week screening period to determine eligibility for study entry. At week 0, volunteers who meet the eligibility requirements will be randomized in a 1:1 ratio to the active control group (8-week, 2 hours/week of lectures) or mindfulness-based intervention (8-week, 2 hours/week of mindfulness meditation training).

ELIGIBILITY:
Inclusion Criteria:

* (1) Brazilian male or female aged between 23 and 65 years and (2) currently working in the classroom

Exclusion Criteria:

1. clinical diagnosis of depression
2. clinical diagnosis of anxiety disorders
3. clinical diagnosis of schizophrenia
4. report of an infectious condition in the last 15 days before collecting a blood sample;
5. had previously practiced or currently practicing meditation, yoga or Tai-Chi.

Ages: 23 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Perceived Stress on the Perceived Stress Scale (PSS-10) at 8-weeks | Baseline and Post-intervention (after 8 weeks)
  Perceived Stress Scale is a validated instrument designed to evaluate the level of subjectively noticed stress, composed of 10 items, 6 of which scoring positively, and 4 scoring negatively, using a Likert-kind frequency scale. The answers range from "Never" (0) to "Always" (4), and the scoring show a crescendo proportional to the experimented stress (0-7 indicating very low stress; 8-11, low stress; 12-15 require attention, 16-20, high stress; above 21, very high stress.
Change from Baseline in Phycological Well-being on the Psychological Well-being Scale (SWB) at 8-weeks | Baseline and Post-intervention (after 8 weeks)
  The 42-item Psychological Wellbeing (PWB) Scale is a validated instrument designed to measures six aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate how strongly they agree or disagree with 42 statements using a 7-point scale (1 = strongly agree; 7 = strongly disagree)
Change from Baseline in DNA methylation at 8-weeks. | Baseline and Post-intervention (after 8 weeks)
  DNA methylation analysis will be performed in blood samples from participants. DNA will be extracted from blood samples and genomic DNA will be converted using EZ® DNA Methylation Gold Kit (Zymo Research, Irvine, CA.) according to the manufacturer's recommendations. Methylation analysis by pyrosequencing of bisulfite-treated genomic DNA was performed by PSQ96ID Pyrosequencer (Qiagen®, Valencia, CA) with reagents PyroMark Gold Q96 (Qiagen®, Valencia, CA) according to the manufacturer's protocol.
Change from Baseline in inflammatory cytokines at 8-weeks. | Baseline and Post-intervention (after 8 weeks)
  Serum samples were obtained through the collection of peripheral blood of the participants. The level of the inflammatory cytokines interleukin-8 (IL-8) pg/mL, interleukin-1β (IL-1β) pg/mL, interleukin-6 (IL-6) pg/mL, interleukin-10 (IL-10) pg/mL, tumor necrosis factor (TNF) pg/mLe interleukin-12p70 (IL-12p70) pg/mL was determined using the Cytometric Bead Array (CBA) Human Inflammatory Cytokines Kit (BD Biosciences, San Jose, CA) and flow cytometry using the FACSCanto II (BD Biosciences, San Jose, CA) cytometer.
Change from Baseline in Cognitive function at 8-weeks. | Baseline and Post-intervention (after 8 weeks)
  Three different neuropsychological tests will be used to evaluate the cognitive function as know:
  1. Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological validated test to assess verbal learning and memory, an assessment of verbal learning over 5 trials, and 30-minute delayed free recall. The test will be applied according to the validation guideline's recommendations.
  2. Trail Making Test (TMT) is a neuropsychological validated test access frontal executive function. The test consists of two parts; the TMT A is a test of visual search and motor speed, whereas the TMT B measures cognitive flexibility, divided attention, and working memory. The test will be applied according to the validation guideline's recommendations.
  3. Stroop Color-Word Test is a validated test used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus. The test comprised four white cards, each 14 × 21.5 cm in size.

SECONDARY OUTCOMES:
Change from Baseline in Positive affect and negative affect at 8-weeks. | Baseline and Post-intervention (after 8 weeks)
  The Positive affect and negative affect scale (PANAS) is evaluate the predominance of positive and negative affects within one's emotional landscape, measures are collected from a 0 ("not a bit") up to 5 ("extremely") range of answers to 20 questions, 10 of which versing about positive affects and dispositions, and 10 about negative emotions and dispositions
Change from Baseline in resilience at 8-weeks. | Baseline and Post-intervention (after 8 weeks)
  The Connor-Davidson Resilience Rating Scale ( CD-RISC )is a 25-item measure of resilience. Each item ranges from 0 ("not true at all") up to 4 ("true nearly all the time"). The final scores are obtained by summing the response to each of the items, with higher values indicating higher levels of resilience
Change from Baseline in sleep quality of at 8-weeks. | Baseline and Post-intervention (after 8 weeks)
  The Pittsburgh Sleep Quality Index (PSQI) provides a subjective measure of sleep quality and patterns.PSQI, a self-administered questionnaire, includes four open-ended questions and 14 questions to be answered using event-frequency and semantic scales. (The latter use paired words of opposite meaning, such as good-bad.) The tool looks at seven areas: subjective sleep quality, sleep latency (the time it takes to fall asleep), sleep duration, habitual sleep efficiency (the ratio of total sleep time to time in bed), sleep disturbances, the use of sleep-promoting medication (prescribed or over-the-counter), and daytime dysfunction.The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Daniela Rodrigues de Oliveira, São Paulo, Brazil